CLINICAL TRIAL: NCT06898528
Title: The Title Used in the Study Protocol: Professor
Brief Title: A Novel Mat Exercise Program Improves Functional Fitness, Activity Levels, and Quality of Life in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen Ching Huang, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C112161; NSTC (Other: National Science and Technology Council)
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Quality of Life; Functional Fitness
Keywords: Exercise game; Functional Fitness; Sport Technology; Physical activity; Stampede training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In this study, investigator recruited older adults aged 60 to 80 years from Taipei City and utilized a parallel experimental design. A total of 32 participants were randomly assigned to either the experimental or control group. A pre- and post-intervention design was implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The implementation of novel exercise mat training program (Experimental): The mat-based exercise facility (Stampede, Taipei, Taiwan) assists participants in exercise training by incorporating interactive light and sound effects to guide users through various exercises while progressively increasing intensity.Participants were randomly assigned to either the experimental or control group. The experimental group underwent a 10-week-long exercise game-based mat training, consisting of two sessions per week (70 min/session), using group-based exercise training.
  Interventions: Behavioral: The group-based mat exercise training on experimental group.
- Active control (Active Comparator): The control group maintained their usual daily activities as active comparator.
  Interventions: Behavioral: The control group

INTERVENTIONS:
Behavioral: The group-based mat exercise training on experimental group. — The training program is divided into two phases: the first phase focuses on fundamental movements, whereas the second phase introduces more advanced exercises. With progress, additional exercise equipment is incorporated, along with increased sets, duration, movement variations, and training intensity. Training sessions (10-week duration) can be conducted in a simple, progressive manner or a game-competitive format.The control group maintained their usual daily activities.
  Arms: The implementation of novel exercise mat training program
Behavioral: The control group — The control group maintained their usual daily activities.
  Arms: Active control

SUMMARY:
In this study, investigators recruited older adults aged 60 to 80 years and utilized a parallel experimental design. A total of 32 participants were randomly assigned to either the experimental or control group. The intervention consisted of a 70-min-long exercise game-based mat training session conducted twice weekly for 10 consecutive weeks. Each session included a 10-min warm-up, approximately 45 min of primary training, and a 15-min cool-down and stretching routine. Participants completed the International Physical Activity Questionnaire (IPAQ) and the World Health Organization Quality of Life questionnaire (WHOQOL, Taiwanese Version) before and after the intervention. Additionally, the functional fitness assessment were conducted.

DETAILED DESCRIPTION:
The mat-based exercise facility (Stampede, Taipei, Taiwan) assists participants in exercise training by incorporating interactive light and sound effects to guide users through various exercises while progressively increasing intensity. The training program is divided into two phases: the first phase focuses on fundamental movements, whereas the second phase introduces more advanced exercises. With progress, additional exercise equipment is incorporated, along with increased sets, duration, movement variations, and training intensity. Training sessions can be conducted in a simple, progressive manner or a game-competitive format. Throughout the training, participants wore a heart rate monitor (ALATHEC Obeat1, Taichung, Taiwan) that recorded their exercise intensity and heart rate fluctuations. However, the exercise intensity and frequency were adjusted based on participants' adaptation. This study encompassed five different lighting modes, namely all light on, circle on, four corners, two lines, and diamond. Each mode was paired with different training protocols and movement patterns, supplemented by training equipment, such as medicine balls, resistance bands, and balance pads.

ELIGIBILITY:
Inclusion Criteria:

(i) Elderly individuals (aged 60-80) who have not experienced any muscle or skeletal injuries in the past month and are able to participate in training normally.

(ii) Completion of the Physical Activity Readiness Questionnaire and meeting the conditions for initiating moderate-intensity exercise intervention.

(iii) Ability to comply with the exercise frequency required by this study and travel to and from the training site independently.

Exclusion Criteria:

(i) individuals with severe musculoskeletal disorders, (ii) individuals deemed unsuitable for exercise training based on a Physical Activity Readiness Questionnaire evaluation or psychiatric disorders, and (iii) individuals under medications that may influence study outcomes.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | The evaluation was conducted at baseline and the 11th week time points.
  The questionnaire was applied to evaluate the physical activities. The duration of activity will be converted into metabolic equivalents (METs), with higher MET values indicating a greater level of physical activity.
World Health Organization Quality of Life questionnaire | The evaluation was conducted at baseline and the 11th week time points.
  The questionnaire was applied to evaluate the quality of life. A self-assessment will be conducted for different dimensions of quality of life, with higher values indicating greater satisfaction in that particular dimension.
Senior fitness | The evaluation was conducted at baseline and the 11th week time points.
  The regular physical fitness was evaluated by indicated senior fitness test. This fitness test measures the number of repetitions performed within a specific time frame, with higher values indicating better fitness. However, for dynamic balance, a shorter time indicates better performance.
Functional fitness | The evaluation was conducted at baseline and 11th week time points.
  The functional fitness was evaluated by sport technology-based AFAscan fitness assessment. This fitness test measures the number of repetitions performed within a specific time frame, with higher values indicating better fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ching Huang, Ph.D., Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peng HT, Tien CW, Lin PS, Peng HY, Song CY. Novel Mat Exergaming to Improve the Physical Performance, Cognitive Function, and Dual-Task Walking and Decrease the Fall Risk of Community-Dwelling Older Adults. Front Psychol. 2020 Jul 24;11:1620. doi: 10.3389/fpsyg.2020.01620. eCollection 2020. PMID 32793044

DOCUMENTS (1):
  • Study Protocol (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT06898528/Prot_000.pdf